CLINICAL TRIAL: NCT00855608
Title: The Safety and Tolerability of Intravitreal Adalimumab in Patients With Refractory Diabetic Macular Retinopathy or Choroidal Neovascularization or Uveitis: A Pilot Study
Brief Title: Intravitreal Adalimumab in Refractory Diabetic Retinopathy, Choroidal Neovascularization or Uveitis: A Pilot Study
Acronym: ADA01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rafic Hariri University Hospital (Other)
Collaborators: American University of Beirut Medical Center (Other)
Responsible Party: Professor Ahmad Mansour, RHUH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHUH
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-09

CONDITIONS: Uveitis; Diabetic Retinopathy; Choroidal Neovascularization
Keywords: choroidal neovascularization; diabetic retinopathy; uveitis; refractory cases of uveitis
MeSH Terms: conditions — Uveitis; Diabetic Retinopathy; Choroidal Neovascularization | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adalimumab arm (Experimental): intravitreal mode of delivery
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — intravitreal adalimumab injection 0.03 ml in volume (1.5mg) one dose to one eye
  Other Names: Humira

SUMMARY:
Direct intravitreal administration of medication is the preferred method of treatment for uveitis and retinal vascular disorders. The eye is a self contained organ relatively isolated from the systemic circulation by the tight blood retinal barrier. Effective intraocular drug levels can be achieved with a much smaller amount of medication if injected intravitreally and this also results in minimal systemic exposure to the patient. Preliminary studies have shown that adalimumab may have a positive role in the management of uveitis in humans and can be an effective treatment intravitreally in animal models. No data has been published yet on intravitreal use of adalimumab in human subjects.

DETAILED DESCRIPTION:
Abstract Purpose: Our aim is study to determine the efficacy and safety of intravitreal adalimumab in patients with active vision threatening uveitis, diabetic macular edema (DME) and choroidal neovascularization (CNV) despite standard treatment and to ensure its safety in intravitreal use in humans and its rapid onset of action.

Design: Pilot study, Non-Randomized, Open Label, Single Group Assignment, Safety Study.

Participants: 15 eyes with refractory CNV, DME, or uveitis will be injected with intravitreal adalimumab on a 3 week interval. Patients will satisfy the inclusion and exclusion criteria listed at the end.

Methods: Initial treatment will consist of intravitreal adalimumab injection (1.5 mg/ 0.03 mL) in the eyes of patients with refractory CNV, DME, or uveitis and with visual acuity less than or equal to 20/70. Patients will be followed up every 3 weeks for a total of 6 weeks. Patients will have a baseline best-corrected visual acuity (BCVA), slit lamp examination, dilated fundus examination, ocular coherence tomography (OCT), fluorescein angiography (F.A), and standard electroretinogram (ERG) and then these studies will be repeated every visit. If there is stabilization or improvement in visual acuity, decrease in edema on OCT and leakage on F.A after the first injection, then further injections will be given. The injection will be delayed if a patient develops an acute systemic infection and will be given when it subsides. If there is worsening of visual acuity after the first injection, patients will be shifted to the traditional treatment with intravitreal Avastin or intravitreal steroids. The paired sample Student t- test, Chi-square test, Pearson correlation and ANOVA will be used to analyze the mean visual acuity and central retinal thickness before and after treatment.

Main outcome measures: to study the response to intravitreal adalimumab injection of patients with different visual acuity at baseline measured in terms of improvement in visual acuity, shrinkage in central retinal thickness, reduction in fluid leakage, and decrease in the active inflammatory uveitis.

Conclusion: Our goal is to study the efficacy and intraocular safety of intravitreal adalimumab in the treatment of refractory CNV, DME, or uveitis.

Background and Significance Inflammatory mediators are involved in the pathogenesis of diabetic retinopathy, choroidal neovascularization and uveitis. Owing to the propensity for visual loss, immunosuppressive treatment in the form of systemic and/or local therapy is often required for the management of cystoids macular edema from posterior uveitis, diabetes or age-related macular degeneration. There have been changes in the management of these conditions over the last few years, with immunomodulatory agents and new intraocular delivery systems. After the new trend of intravitreal corticosteroid and anti-VEGF, the new wave of so-called biologic response modifiers, predominantly monoclonal antibodies directed against inflammatory mediators or their receptors, but also some cytokines, represent a very promising generation of immunomodulating agents. There is rising evidence that these biologic drugs might be superior regarding their anti-inflammatory potential to conventional immunosuppressive therapies. Unfortunately, these new drugs are also very expensive so far. The yearly cost for a regular weight patient is around 20,000 dollars for Adalimumab or Infliximab. Therefore, they may not be universally available in countries with poorly funded health systems and for individuals with low economic status.

Intravitreal injections of anti-VEGF and corticosteroids are currently the standard therapy in a multitude of retinal diseases such as choroidal neovascularization, diabetic maculopathy, proliferative diabetic retinopathy, and uveitis. However many patients respond only partially or develop complications like corticosteroid induced glaucoma or cataract. As such, we are looking for safe new therapies for various chorioretinal disorders aiming at visual improvement.

Adalimumab (Humira) is a genetically engineered antibody against a proinflammatory cytokine, namely, tumor necrosis factor alpha (TNF-α). Adalimumab is the first member of a new class of TNF antibody compounds developed to contain exclusively human sequences. Adalimumab (ADA) is a subcutaneously (SC) self-administered fully human Ig G1 monoclonal antibody directed against tumor necrosis factor alpha (TNFα) which will be used intravitreally.

We do not know if adalimumab injections into the eye are effective and safe in most people. We are performing this pilot study to determine its efficacy and safety in patients with active vision threatening uveitis despite standard immunosuppressive therapy.

Unlike infliximab, adalimumab contains no nonhuman sequences, making it indistinguishable in structure and function from naturally occurring human IgG1. Unlike infliximab, allergic reactions to adalimumab appear to be rare.

Subcutaneous Adalimumab is currently used for the treatment of systemic inflammatory conditions and inflammatory disease of the eye with a relatively favorable safety profile. However, systemic administration carries the risk of systemic side effects, which in the case of adalimumab can be severe, such as increased risk of infection, reactivation of tuberculosis or increased risk for lymphoma.

Intravitreal injection of Adalimumab The eye to be treated will be prepared with 5% povidone-iodine solution after which 1% lidocaine will be administered as a subconjunctival injection about 3 to 4 mm from the limbus to form a small bleb where the intravitreal injection will be given. Following that, 0.03ml of adalimumab will be injected intravitreally using a 30 gauge needle through the pars plana 3.5 mm from the limbus. Twenty minutes after the injection, a paracentesis will be performed in case the intraocular pressure was greater than 25 mmHg or if the optic nerve head was not adequately perfused. By the end of the procedure, the eyes will be covered by a patch for one day after which topical antibiotics (Ciloxan) will be applied 3 times per day for 3 days.

Potential risks Intravitreal adalimumab have never been tried but as any intravitreal intervention, the risks of anti-VEGF therapy consist of local complications including endophthalmitis (0.16% per injection), retinal detachment (0.08% per injection), cataract (0.07% per injection), subconjuntival hemorrhage mainly related to the size of the needle used, and uveitis (0.09% per injection). Systemic administration carries the risk of systemic side effects, which in the case of adalimumab can be severe, such as increased risk of infection, reactivation of tuberculosis or increased risk for lymphoma. However, because the eye is a self contained organ relatively isolated from the systemic circulation by the tight blood retinal barrier, it is unknown how much the amount of the drug injected intravitreally gets reabsorbed systemically.

Post-injection follow-up Patients will be examined every 3 weeks to measure the BCVA along with slit-lamp examination of the anterior segment, dilated fundus examination, OCT, F.A, and ERG. If any of the patients develops a decrease in visual acuity at least five letters of vision post first injection, he/she will be shifted to the traditional treatment with intravitreal avastin or intravitreal steroids. Else, if the vision is stable, patients will continue treatment

The total follow-up period of every patient will be 6 weeks.

Main outcome Our goal is to study the efficacy and intraocular safety of intravitreal adalimumab in the treatment of refractory CNV, DME, or uveitis and to ensure its rapid onset of action. The main outcome measure will be the proportion of patients who lose fewer than 15 letters (3 lines) in BCVA score at 6 weeks compared with baseline. Secondary visual acuity endpoints at 6 weeks include 1) mean change from baseline in BCVA score; 2) the proportion of patients who gain ≥15 letters in BCVA; and 3) the proportion of patients with a Snellen visual acuity of 20/70 or worse compared with baseline. Other secondary endpoints include the effect of adalimumab on the central retinal thickness (CRT) as assessed by OCT and on the lesion size assessed by F.A.

Literature Cited 1-Intravitreal Adalimumab

1A- Manzano et al evaluated the ocular toxicity of escalating doses of intravitreous adalimumab (Humira) in the rabbit eye. Slit-lamp biomicroscopy and fundoscopy were carried out at baseline, day 1, 7 and 14 following intravitreous injection. Escalating doses of intravitreous adalimumab in rabbit eyes caused no detectable functional or structural ocular toxicity up to a dose of 0.50 mg. Administration of 1.0 mg in 0.1 ml was associated with an inflammatory reaction. (Manzano RP et al Ocular toxicity of intravitreous adalimumab (Humira) in the rabbit. Graefes Arch Clin Exp Ophthalmol. 2008 Jun;246(6):907-11).

1B- Use of intravitreal etanercept, another TNF antagonist in humans, with improvement in vision in diabetic macular edema (Tsilimbaris MK,et al. The use of intravitreal etanercept in diabetic macular oedema Semin Ophthalmol 2007 Apr-Jun;22(2):75-9).

1C-Intravitreal Administration of the Anti-Tumor Necrosis Factor Agent Infliximab for Neovascular Age-related Macular Degeneration.Theodossiadis PG, Liarakos VS, Sfikakis PP, Vergados IA, Theodossiadis GP.Am J Ophthalmol. 2009 Feb 9. [Epub ahead of print]

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 17 years
* Patients with active choroidal neovascularization, diabetic retinopathy, or uveitis in the study eye which did not improve with conventional therapy
* Best corrected visual acuity of 20/70 or less.

Exclusion Criteria:

* Are participating in another clinical study requiring follow up examinations
* Have received any other experimental drug within 12 weeks prior to enrollment
* Are unwilling or unable to follow or comply with all study-related procedures
* Inability to obtain photographs, fluorescein angiography, or optical coherence tomography to document CNV, e.g. due to media opacity, allergy to fluorescein dye or lack of venous access
* Aphakia or pseudophakia with the absence of posterior capsule (unless it resulted from a yttrium aluminum garner [YAG]) posterior capsulotomy)
* Within two months prior to screening, have had intraocular surgery (including cataract surgery) in the study eye
* Within 1 month prior to screening had YAG laser in the study eye
* Have had intravitreal anti VEGF or intravitreal steroids in the last 6 weeks
* Have had previous pars plana vitrectomy in the study eye
* Are pregnant or are trying to become pregnant
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated

Ages: 17 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The main outcome measure will be visual acuity improvement (3 lines) | 6 weeks

SECONDARY OUTCOMES:
central foveal thickness and angiographic lesion size | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ahmad m mansour, md, Principal Investigator — RHUH
Locations (1):
- Rafic Hariri University Hospital, Beirut, South Beirut, Lebanon

REFERENCES:
- [Result] Theodossiadis PG, Liarakos VS, Sfikakis PP, Vergados IA, Theodossiadis GP. Intravitreal administration of the anti-tumor necrosis factor agent infliximab for neovascular age-related macular degeneration. Am J Ophthalmol. 2009 May;147(5):825-30, 830.e1. doi: 10.1016/j.ajo.2008.12.004. Epub 2009 Feb 10. PMID 19211094